CLINICAL TRIAL: NCT01261104
Title: Relationship Between Hearing Thresholds, Handicap and Time for Treatment-seeking in a Public Hearing Healthcare Service
Brief Title: Relationship Between Hearing Thresholds, Handicap and Time for Treatment-seeking
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Deborah Viviane Ferrari, Professor, Faculdade de Odontologia de Bauru
Other Study IDs: FOBCEP104/2010
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Hearing Impairment
Keywords: hearing loss; handicap; counseling
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hearing impaired elderly
- Hearing impaired adults

SUMMARY:
Purpose: to investigate the relationship between time for treatment seeking and audiometric data and self-assessment of handicap for patients in a public hearing healthcare service. Methods: Retrospective study. Records of 152 elderly and 48 adults with hearing impairment were analyzed. The ISO audiometric thresholds average (500 to 4000Hz) and high frequencies average (2000 to 6000Hz), the speech recognition thresholds and the total, social and emotional scores from the Hearing Handicap Inventory for the Adults (HHIA) and Elderly (HHIE) were compared with the time between the onset of hearing complaints and the first treatment seeking. Results: The average time for treatment seeking was 7,6 years. No statistical difference was found between ISO and high frequency audiometric average, HHIA/E scores and time for treatment seeking between adults and the elderly. Weak but significant negative correlations were observed between the audiometric data and time for treatment seeking. There was no relationship between the time for treatment seeking and educational, socioeconomic levels and perception of handicap. Conclusions: The search for treatment seems to be multifactorial. Despite technological advances and changes in access to information and treatment time for treatment seeking was similar to that reported 30 years ago.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old. Without experience with hearing aid use. Diagnosed with sensorineural hearing loss. Audiogram data available

Exclusion Criteria:

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hearing impaired adults and elderly attended at a public hearing healthcare service
Sampling Method: Non-Probability Sample
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Ferrari, PhD, Principal Investigator — Faculdade de Odontologia de Bauru
Locations (1):
- Faculdade de Odontologia de Bauru, Bauru, São Paulo, Brazil